CLINICAL TRIAL: NCT05841303
Title: Comparative Evaluation of Vitamin C and Injectable-platelet Rich Fibrin in the Management of Thin Gingival Phenotype: A Split-mouth Randomized Clinical Trial.
Brief Title: Comparative Evaluation of Vitamin C and Injectable-platelet Rich Fibrin in the Management of Thin Gingival Phenotype
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Mahmoud Mohamed Mohamed Abdelhay, Teaching assistant at periodontology department MTI University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13123PER 3_3_1
Record Dates: First submitted 2023-04-07; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Thin Gingival Biotype
Keywords: Thin gingival biotype; Vitamin C; i-PRF; Microneedle
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: A Split-mouth Randomized Clinical Trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each site with thin gingival phenotype will be randomly allocated to either intervention group (vit. C with MN) or control group (I-PRF with MN). The allocation sequence will be concealed in opaque sealed envelopes, which will be identified with the initials of the patient's name. For each patient, the envelope will be opened immediately before the intervention. Patients will be blinded during the intervention and follow-up sessions.
  * The patients will be blinded
  * The operator will be blinded as investigator can give the operator the vial filled with either
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vit. C injection (Experimental): Derma pen device model M8 with 24 -micro needle will be adjusted with 1.5 mm depth at the 6th mode speed of 700 cycles/min with intermittent motion used on the sextant gingival area for 30-40 seconds/tooth.
  vitamin C will be injected with microneedle at two points for each site in the attached gingiva of one site of the jaw either the left or the right side at 3 mm apical to the free gingival margin in the facial side of the tooth until the blanching of the gingiva will be seen and apical to the mucogingival junction.
  - Vitamin C will again be injected at the same site after 1 week and after 2 weeks from the baseline final injection which will be given.
  Interventions: Drug: Vit C
- Injectable-platelet Rich Fibrin (i-PRF) (Active Comparator): The derma pen will be used same as vitamin C group. I-PRF will be immediately aspirated using micro needle. I-PRF will be injected on the site with thin gingival phenotype (split mouth technique) with micro needling with derma pen at two points for each site in the attached gingiva at 3 mm apical to the free gingival margin in the facial side of the tooth until the blanching of the gingiva was seen and apical to the mucogingival junction.
  4. I-PRF will again be injected at the same site after 1 week and after 2 weeks from the baseline final injection which will be given.
  Interventions: Other: injectable PRF

INTERVENTIONS:
Drug: Vit C — Vit c is proven to be an anti-inflammatory and antioxidant agent. also play a great role in collagen biosynthesis (collagen type I), as it helps in fibroblasts proliferation. It reduces the potentiality of scaring via inhibiting cross-linking of collagen fibers and fibrosis. It acts as a cofactor in hydroxyproline synthesis to produce collagen type IV and improves endothelial cell vitality and function..
  Other Names: Ascorbic acid
  Arms: Vit. C injection
Other: injectable PRF — 5 ml of peripheral blood from each patient , blood will be transferred to a glass coated plastic vacutainer tube without anticoagulant. Then this tube will immediately centrifuged at 700 rpm for 3 mins [Centrifuge Machine 5000rpm.After centrifugation, two fluid layers will formed, upper being yellow fluid layer (i-PRF) while lower layer containing red blood cells. Yellow fluid layer containing i-PRF will be immediately aspirated using micro needle to be injected for management of gingival phenotype
  Other Names: i-PRF
  Arms: Injectable-platelet Rich Fibrin (i-PRF)

SUMMARY:
* The goal is to compare between the effect of vitamin C and Injectable-platelet rich fibrin in the management of thin gingival phenotype.
* The main question: ln patients with thin phenotype, will injecting Vitamin C with micro needles increase the gingival thickness compared to injecting injectable-platelet rich fibrin with micro needles?

  * After enrolment, periodontal examination and measurement of periodontal probing depth (PD), patients with a high periodontal probe visibility in the anterior teeth will be identified. These patients will undergo gingival thickness (GT) measurement using trans gingival probing technique in the anterior teeth, and those with a measured GT of ≤ 1.5mm will be diagnosed with thin phenotype.
  * Keratinized tissue width will be measured.
* Micro needle the gingival mucosa by using derma pen device which will be used in intermittent motion on the sextant gingival area for 30-40 seconds/tooth. When bleeding pinpoints observed on all areas of attached gingiva.

  * Intervention group: Vitamin C injection will be injected with microneedle at two points for each site in the attached gingiva of right or left (split mouth) at 3 mm apical to the free gingival margin in the facial side of the tooth until the blanching of the gingiva will be seen and apical to the mucogingival junction.
  * Control group:

    1.Preparation and administration of injectable platelets rich fibrin (i-PRF). I-PRF will be injected on the site with thin gingival phenotype on the other side of the jaw in the same patient (split mouth technique) with micro needling same way as vitamin C group.

    3.Vitamin C and I-PRF will again be injected at the same site after 1 week and after 2 weeks from the baseline final injection which will be given.

Outcomes: The results for the mean gingival thickness (GT), keratinized tissue width (kTW), pocket depth (PD), and gingival index (GI) at baseline, 1 month, 3 months and after 6 months

DETAILED DESCRIPTION:
Research objective: The aim of conducting this research is development of newer, less invasive therapeutic approaches that help in prevention of gingival recession. As thin gingival biotype is more prone to gingival recession and to achieve satisfactory therapeutic results with minimum trauma to tissues of any interventional process.

Research Procedure in brief:

This study will be carried out on patients enrolled from the Outpatient Clinic of Oral Medicine and Periodontology department, Faculty of Dentistry, Cairo University.

General operative procedures

* The patients who fulfil the inclusion criteria will be enrolled. The nature of the study will be explained to each patient as well as the importance of compliance with pre- and post-operative instructions and follow-up visits.
* Each patient will be asked to sign an informed consent (appendix 1)
* After enrolment, periodontal examination and measurement of periodontal probing depth (PD), patients with a high periodontal probe visibility in the anterior teeth will be identified. These patients will undergo gingival thickness (GT) measurement using trans gingival probing technique in the anterior teeth, and those with a measured GT of ≤ 1.5mm will be diagnosed with thin phenotype.
* The methods used for evaluation of gingival thickness included Visual assessment with aid of probe and direct measurement by #15 endodontic spreader will be inserted trans gingivally into the anaesthetized selected site (anaesthetized with Lidocaine 10% spray), stopper will be used as the reference point and the exact measurement will be recorded with the help of endo-ruler or caliber.
* Keratinized tissue width will be measured from gingival margin to mucogingival junction with the help of calibrated periodontal probe (UNC 15 probe).
* As a preliminary routine, supragingival scaling will be performed and oral hygiene instructions will be provided by the dental hygienist. We subsequently will schedule the procedure and perform it aseptically.
* The area to be injected will be anesthetized. To microneedle the gingival mucosa, we will use a derma pen device model M8 with 24 microneedles arranged in rows, which will be adjusted with 1.5 mm depth at the 6th mode speed of 700 cycles/min. The derma pen will be used in intermittent motion on the sextant gingival area for 30-40 seconds/tooth. When bleeding pinpoints observed on all areas of attached gingiva, the gingival mucosa will be irrigated with a saline solution and sterile gauze will be applied to dry the area.
* Intervention group: Vitamin C injection will be injected with microneedle at two points for each site in the attached gingiva of one site of the jaw either the left or the right side and the other side will be injected with injectable platelets rich fibrin (i-PRF) as a control group at 3 mm apical to the free gingival margin in the facial side of the tooth until the blanching of the gingiva will be seen and apical to the mucogingival junction. The treated area will be left without dressing. The patient will be instructed to refrain from drinking acidic or hot beverages for 24 hours and to not brush the teeth of the injected area for one day to avoid any mechanical trauma to the gingiva. Following the procedure, neither mouthwashes nor medications will be prescribed.
* Control group:

  1. Preparation and administration of injectable platelets rich fibrin (i-PRF): After collection of 5 ml of peripheral blood from each patient, blood will be transferred to a glass coated plastic vacutainer tube without anticoagulant. Then this tube will immediately centrifuged at 700 rpm for 3 mins [Centrifuge Machine 5000rpm]. After centrifugation, two fluid layers will formed, upper being yellow fluid layer (i-PRF) while lower layer containing red blood cells. Yellow fluid layer containing i-PRF will be immediately aspirated using micro needle.
  2. I-PRF will be injected on the site with thin gingival phenotype on the other side of the jaw in the same patient (split mouth technique) with micro needling with derma pen at two points for each site in the attached gingiva at 3 mm apical to the free gingival margin in the facial side of the tooth until the blanching of the gingiva was seen and apical to the mucogingival junction.
  3. Vitamin C and I-PRF will again be injected at the same site after 1 week and after 2 weeks from the baseline final injection which will be given.

Outcomes: The results for the mean gingival thickness (GT), keratinized tissue width (kTW), pocket depth (PD), and gingival index (GI) at baseline, 1 month, 3 months and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy individuals of age ≥ 18 to 40 years with absence of active periodontal disease.

* Having thin gingival phenotype <1.5mm.
* No systemic disease according to Modified Cornell Medical Index health questionnaire.
* Non-smoker.
* Full mouth plaque index (PI) and full-mouth bleeding on probing (BOP) score of ≤ 15%.
* No malocclusion, crowding, fillings, missing or supernumerary mandibular anterior teeth.
* No blood-borne conditions.

Exclusion Criteria:

* Active orthodontic treatment.
* Previous periodontal surgery.
* Systemic disease.
* Use of blood thinners.
* Use of any drugs that might lead to gingival enlargement.
* Mucogingival stress, bruxism.
* Pregnancy or lactation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Gingival thickness (GT) change from baseline to 6months. | GT will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  GT will be measured using a no. 15 endodontic spreader (the file will be inserted perpendicularly through the gingiva, 2 mm apical to the gingival margin through the soft tissue until a hard surface reached). The flowable light-curing composite will be used to mark the penetration thickness on the spreader. Then, caliper or endo. Ruler will be used to measure the penetration thickness between the spreader's tip and the light-cured composite.

SECONDARY OUTCOMES:
Keratinized tissue width (KTW) change from baseline to 6months. | The KTW. will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  The KTW will be calculated from the gingival margin to the mucogingival junctions with the help of a periodontal probe (UNC-15).
Gingival index (GI)change from baseline to 6months. | GI. will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  The GI is used to assess the gingival condition based on the following criteria 0=normal gingiva.
  1. mild inflammation (slight change in color and slight edema but no BOP).
  2. moderate inflammation (redness, edema, and glazing, bleeding on probing).
  3. severe inflammation (marked redness and edema, ulceration with tendency to spontaneous bleeding).
  The scores of the four areas of the tooth (buccal, mesial, distal, lingual) can be summed and divided by four to give the GI for the tooth.
Plaque index (PI) change from baseline to 6months. | PI will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  PI will be measured using UNC periodontal probe at six sites per tooth.
Probing depth. (PD) change from baseline to 6months. | PD. will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  PD will be measured from the gingival margin to the bottom of the gingival sulcus/ periodontal pocket using UNC periodontal probe at six sites per tooth

CONTACTS AND LOCATIONS:
Overall Officials: Riham M. Omar, Professor, Study Director — Cairo University
Locations (1):
- Faculty of dentistry Cairo University, Cairo, Elmanil, Egypt